CLINICAL TRIAL: NCT02290366
Title: Prospective Evaluation of Focal Brachytherapy Using Cesium-131 For Patients With Low Risk Prostate Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator decision
Sponsor: Ronald M. Benoit, MD (Other)
Responsible Party: Sponsor-Investigator, Ronald M. Benoit, MD, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO14020322
Record Dates: First submitted 2014-11-05; First posted 2014-11-14 (Estimated); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Cesium-131

STUDY DESIGN:
Intervention Model Description: Brachytherapy, using Cesium 131
Oversight: Data Monitoring Committee: No

ARMS (1):
- Focal Therapy (Experimental)
  Interventions: Radiation: Focal prostate brachytherapy with Cesium-131

INTERVENTIONS:
Radiation: Focal prostate brachytherapy with Cesium-131

SUMMARY:
The standard options for men with very low risk prostate cancer include active surveillance and the standard treatment options for low risk disease, i.e. radical prostatectomy, external beam radiotherapy, and whole gland prostate brachytherapy. The present study seeks to evaluate focal brachytherapy using the isotope Cesium 131 to treat patients with low risk prostate cancer. The goals of the study are to determine the biochemical disease free survival at five years in these patients, as well as to determine the acute and late urinary, bowel, and sexual toxicity associated with focal prostate brachytherapy using Cesium 131. Patients eligible for the study will be men with histologically confirmed adenocarcinoma of the prostate with clinical stage T1c-T2aN0M0, Gleason score ≤3+3=6, prostate specific antigen(PSA) <10 ng/ml or a PSA density ≤ 0.15 ng/cc, and ≤ 2 cores positive out of a minimum of 12 cores sampled. Additionally, patients must have a single, dominant index lesion on MRI. The study is a phase II study. Patients will be followed prospectively. Dosimetry will be evaluated post-procedure, and PSAs will be obtained every three months in year one and every six months from year two through year five. Urinary, bowel, and sexual morbidity will be assessed by patient survey prior to treatment , two weeks, after treatment, at three month intervals in year one and at six month intervals in years two through five.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate
* Clinical stage T1c-T2aN0M0
* Gleason score <= 3+3=6
* prostate specific antigen (PSA) <10 ng/ml
* <= 2 cores positive out of a minimum of 12 cores sampled

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
biochemical disease free survival | five years

CONTACTS AND LOCATIONS:
Locations (1):
- UPMC Mercy, Pittsburgh, Pennsylvania, United States